CLINICAL TRIAL: NCT01890993
Title: Retrospective Collection of Effectiveness and Safety Data From Patients Treated With Liraglutide or DPP-4 Inhibitor in Primary Care in Europe
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4077; U1111-1142-2764 (Other: WHO); ENCEPP/SDPP/8135 (Other: EU PAS)
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Liraglutide
  Interventions: Drug: liraglutide
- DPP-4
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Anonymised patient level data will be collected by the patients' own general practitioner and electronic case report form (eCRF) will be used to capture the data.

SUMMARY:
This study is conducted in Europe. The aim of this study is to demonstrate the clinical effectiveness and safety of liraglutide and dipeptidyl peptidase-4 (DPP-4) inhibitor therapy in routine primary care in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with liraglutide or DPP-4 inhibitors, according to license in respective participating country with data available for 12 (+/- 2) months

Exclusion Criteria:

* Patients treated with liraglutide or DPP-4 inhibitors, outside of license in respective participating country

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with type 2 diabetes initiated on liraglutide or a DPP-4 inhibitor and primarily managed in primary care with 12 (+/-2) months of available data will be included in this study. Only data derived from patients receiving either therapy in accordance with license indications will be included and analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated haemoglobin) | Baseline (anytime within 3 months before therapy initiation), month 12 (+/-2)

SECONDARY OUTCOMES:
Change in body weight | Baseline (anytime within 3 months before therapy initiation), month 12 (+/-2)
Change in systolic blood pressure | Baseline (anytime within 3 months before therapy initiation), month 12 (+/-2)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Paris La Défense Cedex, France
- Mainz, Germany
- Madrid, Spain
- Crawley, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com